CLINICAL TRIAL: NCT03540017
Title: A Pilot Study of Heated Intraperitoneal Chemotherapy (HIPEC) After Interval Cytoreductive Surgery (CRS) in Patients Who Have Received Neoadjuvant Chemotherapy (NACT) for Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancers
Brief Title: HIPEC After Initial CRS in Patients Who Have Received NACT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Collaborators: Katie Oppo Research Fund (Unknown)
Responsible Party: Principal Investigator, Jill Whyte, Physician, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB #: 18-0153
Record Dates: First submitted 2018-04-16; First posted 2018-05-30 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIPEC (Experimental): Patient will receive HIPEC in the form of Cisplatin 100mg/m2. 5. HIPEC will be provided at completion of surgical cytoreduction. The chemotherapy will be ordered by the treating gynecologic oncologist. It will be prepared in the chemotherapy pharmacy and delivered to the operating room once the surgeon confirms optimal cytoreduction and eligibility. Patients undergoing bowel resection will be left with bowel in discontinuity during the HIPEC infusion cycle. The abdomen will be temporarily closed with skin staples to prevent spillage of the perfusate. HIPEC will be delivered using the closed technique as has been well described.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Heated Intraperitoneal Chemotherapy will be administered after the completion of interval cytoreductive surgery after three cycles of neoadjuvant chemotherapy.

SUMMARY:
The majority of women diagnosed with ovarian, fallopian tube and primary peritoneal cancer present with advanced stage III and IV disease. Despite aggressive surgery and systemic chemotherapy, the majority of patients will relapse. Five year survival remains only 20-35% for patients diagnosed with bulky stage IIIC and IV cancers. Patients who are not candidates for an initial cytoreductive surgery at the time of diagnosis form a particularly poor prognosis group. These patients are treated with neoadjuvant chemotherapy (NACT) and will ultimately undergo cytoreductive surgery provided there is a response to chemotherapy. New therapies for this cohort of women are urgently needed.

The investigators have designed a pilot study to evaluate the feasibility of heated intraoperative peritoneal chemotherapy (HIPEC) given at the time of interval cytoreductive surgery after 3 cycles of NACT. Patients undergoing NACT for ovarian, fallopian tube or primary peritoneal cancer will be evaluated after their third cycle of chemotherapy for trial participation. Patient meeting eligibility criteria will proceed with cytoreductive surgery. HIPEC will be administered in those patients in whom optimal tumor cytoreduction is achieved. Primary objective of this study is to evaluate the feasibility, toxicity and tolerability of HIPEC administered after NACT.

DETAILED DESCRIPTION:
Cancer of the ovary, fallopian tube and peritoneum (referred to as epithelial ovarian cancer, EOC) remains the leading cause of death from gynecologic cancer in the US and is expected to account for 22,000 cases and 14,000 deaths in 2016. Patients classically present with peritoneal carcinomatosis and ascites, a reflection of the dissemination pattern of this cancer in the peritoneal cavity. Malignant cells in EOC disseminate throughout the peritoneal cavity forming tumors on the parietal and visceral peritoneum. The majority of patients will be found to have advanced International Federation of Gynecology and Obstetrics (FIGO) stage III and IV disease at initial presentation. Patients with peritoneal carcinomatosis from EOC most often succumb to advanced locoregional disease in the form of intractable ascites, malignant visceral obstruction and cancer cachexia.

Primary cytoreductive surgery (PCS) followed by systemic chemotherapy has been the standard of care for women presenting with advanced EOC. The ability to achieve optimal surgical cytoreduction is historically the most important prognostic factor for women with EOC. The Gynecologic Oncology Group defines optimal cytoreduction as a post-operative residual disease of ≤ 1 cm in largest diameter . Wide variability in the extent and effort of cytoreductive surgery is seen in clinical practice with surgical cytoreductive efforts ranging from standard procedures (hysterectomy, salpingo-opherectomy, omentectomy) to complex multiviceral resections that may require radical upper abdominal surgery. There is increasing evidence that the patients who ultimately gain the most benefit from surgery are those with no gross residual disease (R0 resection) at the completion of PCS . An examination of 2,655 patients with epithelial ovarian cancer or primary peritoneal cancer enrolled in the Gynecologic Oncology Group 182 study demonstrated improved OS and PFS in those patients with in whom PCS resulted in a complete gross resection . Patients presenting with bulky upper abdominal disease (UAD) have a particularly poor prognosis. Women presenting with bulky UAD have been shown to have inferior PFS and OS survival compared to patents with no or limited UAD even among patients in whom optimal debulking surgery is successfully performed . Importantly, the presence of bulky UAD is associated with diminishing rates of successful PCS.

Advanced stage EOC is heterogenous, ranging from limited intra-abdominal disease to diffuse carcinomatosis involving the majority of the peritoneal surfaces. Use of a universal staging system for peritoneal malignancy may aid the clinician in treatment planning and prognostication. While several attempts have been made to develop peritoneal cancer scoring systems, the most widely used is the Peritoneal Cancer Index (PCI) as described by Jacquet and Sugarbaker in 1996 . The PCI quantitates the volume of tumor implants in 13 different abdomino-pelvic regions which are added up to form a score ranging from 0-39. While the PCI may be used as a prognostic indicator, it does not directly correlate with resectability of the disease. Tumor involvement of critical anatomic sites, for example regions 9, 10 and 11, representing the jejunum and ileum, may be associated with unresectable disease despite a low PCI score .

Two recently published randomized controlled trials demonstrated that neoadjuvant chemotherapy (NACT) and interval cytoreductive surgery (ICS) was non-inferior to PCS and adjuvant chemotherapy and resulted in a lower incidence of treatment related morbidity and mortality. These trials, however, have been criticized for lower optimal debulking rates and significantly lower median overall survival rates compared to prior trials in advanced EOC. The choice between PCS and NACT remains controversial and clinical guidelines have recently been published to aid clinicians in the choice between these treatment plans .

Patients who are not candidates for PCS due to medical comorbidities, poor performance status or clinically apparent or obvious unresectable disease constitute a group with a particularly poor prognosis. These patients are preferentially treated with neoadjuvant chemotherapy (NACT). NACT is associated with decreased peri-operative morbidity and an increased likelihood of optimal cytoreduction at surgery compared with primary surgery, however, to date a survival benefit or improvement has not been demonstrated . A recent multi-institutional observational study evaluating the use of NACT in patients with stage III/IV EOC at 6 NCI designated cancer centers demonstrated a significant increase in the use of NACT since 2010, from 16 - 34% in stage III and from 41 - 62% in stage IV EOC . Patients who received NACT were more likely to undergo optimal CRS but were less likely to require ICU admission or re-hospitalization. Among women with stage IIIC disease who had optimal CRS to ≤1 cm, NACT was associated with decreased overall survival when compared to PCS. This difference in survival, however, did not persist in NACT patients in whom CRS resulted in no gross residual disease.

Because of the tendency for EOC to remain confined within the peritoneal cavity for much of the course of disease, the use of post-operative intra-peritoneal (IP) chemotherapy has been extensively evaluated in women who have undergone successful cytoreductive surgery (CRS). Four large randomized clinical trials have been performed by the Gynecologic Oncology Group (GOG), three of which demonstrate improved overall survival in patients treated with an IP regimen. GOG 172 demonstrated a striking 16 month improvement in overall survival in patient's receiving IP cisplatin and paclitaxel when compared to patients receiving intravenous cisplatin and paclitaxel, a survival difference that was sustained in a follow-up publication after a median 10 year survival . Despite randomized controlled trial (RCT) evidence supporting a survival advantage for IP chemotherapy, its use remains low, largely due to potential toxicity and possible IP catheter complications. Despite optimal CRS and systemic chemotherapy the majority of patients will ultimately experience recurrence of the disease.

Heated intra-operative peritoneal chemotherapy (HIPEC) has garnered interest in the international oncology community for the treatment of peritoneal surface malignancies. HIPEC has demonstrated clinical efficacy for the treatment of pseudomyxoma peritonei, appendiceal cancer, colon cancer and malignant mesothelioma. HIPEC allows for the treatment of residual microscopic disease at the completion of CRS. HIPEC takes advantage of the plasma-peritoneal barrier to allow for peritoneal drug levels 20-1000 times that seen in plasma . HIPEC to >41°C may have anti-tumor effects as well as allow for better penetration of the drug into residual tumor . The use of HIPEC at the time of surgery, prior to the formation of adhesions, may allow for improved distribution of chemotherapy throughout the peritoneal cavity.

HIPEC has been investigated as a treatment for patients with newly diagnosed EOC as well as for patients with recurrent disease. Retrospective and case-control studies show a survival advantage for patients in both the primary and recurrent disease setting.

A recent randomized controlled study performed in Europe was the first well-designed, randomized, prospective clinical trial to demonstrate a survival advantage for HIPEC in EOC . This phase 3 randomized trial evaluated the administration of HIPEC using cisplatin in women undergoing interval cytoreductive surgery after NACT and demonstrated a significant improvement in progression free and overall survival with acceptable toxicity.

By far, the most common drug evaluated in HIPEC for EOC is Cisplatin. Cisplatin (CDDP) is a heavy metal complex containing a central atom of platinum surrounded by two chloride atoms and two ammonia molecules in the cis- position. It has biochemical properties similar to that of bifunctional alkylating agents producing inter- and intra-strand cross-links in DNA. It is non-cell-cycle specific. Approximately 95% of the dose is absorbed from the peritoneal cavity in 1.0 hour. CDDP concentrates in the liver, kidney and intestine and is excreted by the kidneys. The dose of CDDP recommended for normothermic intraperitoneal administration is the same as that recommended for intravenous administration and ranges from 75 -100 mg/m2. The major dose-limiting toxicity of CDDP is dose-related cumulative renal insufficiency. Other toxicities include ototoxicity, myelosuppression, nausea and vomiting, hair loss and peripheral neuropathy.

A recent phase I multicenter trial of NACT followed by HIPEC in EOC using CDDP established a dose of 70 mg/m2 as a tolerable dose in patients who had received 6 cycles of carboplatin and paclitaxel neoadjuvant chemotherapy . The results of this recently published phase I clinical trial are encouraging. However, in current clinical practice, patients tend to receive 3 cycles of NACT with carboplatin and paclitaxel based regimens followed by CRS, as opposed to 6 initial cycles of NACT given in the phase I study.

The investigators propose a pilot study evaluating the feasibility of HIPEC in women undergoing interval CRS and achieving optimal tumor cytoreduction after 3 cycles of NACT. The safety, tolerability and efficacy of HIPEC will be evaluated in this cohort of EOC patients with historically inferior outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed cancer of the ovary, fallopian tube or peritoneum.
2. Women of all races and ethnicities are eligible for this trial.
3. Age > 18.
4. The patient must have documented disease limited to the abdomen and pelvis that is amenable to complete CRS indicated by:

   1. Disease confined to the peritoneal surfaces.
   2. No clinical or radiological evidence of hematogenous or distant (extra-abdominal) nodal metastasis.
5. Evidence of response to NACT must as documented by at least one of the following: decline in serum CA125 level, at least a 30% decrease in the sum of the longest diameter of target lesions on radiographic imaging, or resolution of ascites or pleural effusion(s).
6. Gynecologic Oncology Group (GOG) performance status <= 2
7. Leukocytes >= 3,000/microliter (mcL), absolute neutrophil count >= 1,500/mcL, platelets >= 100,000/mcL
8. Adequate hepatic function as measured by total bilirubin within normal institutional limits, aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x institutional upper limit of normal
9. Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min for patients with creatinine levels above institutional normal
10. Albumin >= 2.5 mg/dL
11. Satisfactory cardiopulmonary function (no history of severe congestive heart failure or severe pulmonary disease, as indicated by clinically acceptable risks to undergo major abdominal surgery
12. Voluntary participation after getting written informed consent

Exclusion Criteria:

1. Prior chemotherapy (other than NACT) or whole abdomen radiation for ovarian, fallopian tube or primary peritoneal cancers.
2. Patients with an active second malignancy regardless of site.
3. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
4. Pregnant or breast-feeding patients
5. Patients who are receiving other oncologic investigational therapeutic agents
6. Patients receiving NACT whose disease has progressed following at least 3 cycles of platinum-based therapy, defined by at least one of the following: clinical deterioration (new or worsening of existing ascites, carcinomatous ileus, malignant bowel obstruction, declining performance status); new lesion(s) or increase in maximal diameter of > 20% of the two largest target lesions; rising CA-125 (an increase of at least 10% of baseline value that increases over 3 values obtained every 21 days).
7. Cardiac or pulmonary conditions that preclude aggressive cytoreductive surgery.
8. Patients found to have non-gynecologic cancer at the time of surgery.
9. Patients with gynecologic malignancy of low-grade serous or borderline histology.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2024-07-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Morbidity, assessed by the occurrence of adverse events and serious adverse events | 30 days
  Severity of adverse events will be evaluated using the NCI Common Terminology Criteria for Adverse Events version 4.0 [NCI CTCAE v4.0]. AEs will be classified as possibly, probably, or definitely related to study treatment.
Safety data obtained from scheduled exams | 1 year
  Physical examinations, vital signs, hematologic and clinical parameters, measured monthly for 12 months after initial study treatment or subject discontinuation, whichever comes first.
Mortality | 5 years
  Time from surgery date to death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Time from surgery date to the first documentation of disease progression or death due to any cause.
Ability to complete systemic IV chemotherapy after IDS and HIPEC | 1 year
  Patient completion of systemic IV chemotherapy after surgery and HIPEC.
Functional Assessment of Cancer Therapy-Ovarian (FACT-O) | 2 years
  Survey administered to assess for quality of life.
Completeness of surgical cytoreduction | 24 hours
  Complete cytoreduction will be determined as having a CC score of 0 or 1
Achievement of hyperthermia | 24 hours
  Target intra-peritoneal temperature of 41-43°C.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Whyte, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang SJ, Hodeib M, Chang J, Bristow RE. Survival impact of complete cytoreduction to no gross residual disease for advanced-stage ovarian cancer: a meta-analysis. Gynecol Oncol. 2013 Sep;130(3):493-8. doi: 10.1016/j.ygyno.2013.05.040. Epub 2013 Jun 6. PMID 23747291
- [Result] Gomez-Hidalgo NR, Martinez-Cannon BA, Nick AM, Lu KH, Sood AK, Coleman RL, Ramirez PT. Predictors of optimal cytoreduction in patients with newly diagnosed advanced-stage epithelial ovarian cancer: Time to incorporate laparoscopic assessment into the standard of care. Gynecol Oncol. 2015 Jun;137(3):553-8. doi: 10.1016/j.ygyno.2015.03.049. Epub 2015 Mar 28. PMID 25827290
- [Result] Horowitz NS, Miller A, Rungruang B, Richard SD, Rodriguez N, Bookman MA, Hamilton CA, Krivak TC, Maxwell GL. Does aggressive surgery improve outcomes? Interaction between preoperative disease burden and complex surgery in patients with advanced-stage ovarian cancer: an analysis of GOG 182. J Clin Oncol. 2015 Mar 10;33(8):937-43. doi: 10.1200/JCO.2014.56.3106. Epub 2015 Feb 9. PMID 25667285
- [Result] Zivanovic O, Sima CS, Iasonos A, Hoskins WJ, Pingle PR, Leitao MM Jr, Sonoda Y, Abu-Rustum NR, Barakat RR, Chi DS. The effect of primary cytoreduction on outcomes of patients with FIGO stage IIIC ovarian cancer stratified by the initial tumor burden in the upper abdomen cephalad to the greater omentum. Gynecol Oncol. 2010 Mar;116(3):351-7. doi: 10.1016/j.ygyno.2009.11.022. PMID 20022092
- [Result] Jacquet P, Sugarbaker PH. Clinical research methodologies in diagnosis and staging of patients with peritoneal carcinomatosis. Cancer Treat Res. 1996;82:359-74. doi: 10.1007/978-1-4613-1247-5_23. PMID 8849962
- [Result] Spiliotis J, Halkia EE, Kalantzi N, Giassas S, Lianos E, Efstathiou E, Sugarbaker PH. Mapping the location of peritoneal metastases using the peritoneal cancer index and the correlation with overall survival: a retrospective study. J BUON. 2015 May;20 Suppl 1:S64-70. PMID 26051335
- [Result] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Result] Kehoe S, Hook J, Nankivell M, Jayson GC, Kitchener H, Lopes T, Luesley D, Perren T, Bannoo S, Mascarenhas M, Dobbs S, Essapen S, Twigg J, Herod J, McCluggage G, Parmar M, Swart AM. Primary chemotherapy versus primary surgery for newly diagnosed advanced ovarian cancer (CHORUS): an open-label, randomised, controlled, non-inferiority trial. Lancet. 2015 Jul 18;386(9990):249-57. doi: 10.1016/S0140-6736(14)62223-6. Epub 2015 May 19. PMID 26002111
- [Result] Wright AA, Bohlke K, Armstrong DK, Bookman MA, Cliby WA, Coleman RL, Dizon DS, Kash JJ, Meyer LA, Moore KN, Olawaiye AB, Oldham J, Salani R, Sparacio D, Tew WP, Vergote I, Edelson MI. Neoadjuvant Chemotherapy for Newly Diagnosed, Advanced Ovarian Cancer: Society of Gynecologic Oncology and American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2016 Oct 1;34(28):3460-73. doi: 10.1200/JCO.2016.68.6907. Epub 2016 Aug 8. PMID 27502591
- [Result] Meyer LA, Cronin AM, Sun CC, Bixel K, Bookman MA, Cristea MC, Griggs JJ, Levenback CF, Burger RA, Mantia-Smaldone G, Matulonis UA, Niland JC, O'Malley DM, Wright AA. Use and Effectiveness of Neoadjuvant Chemotherapy for Treatment of Ovarian Cancer. J Clin Oncol. 2016 Nov 10;34(32):3854-3863. doi: 10.1200/JCO.2016.68.1239. PMID 27601552
- [Result] Alberts DS, Liu PY, Hannigan EV, O'Toole R, Williams SD, Young JA, Franklin EW, Clarke-Pearson DL, Malviya VK, DuBeshter B. Intraperitoneal cisplatin plus intravenous cyclophosphamide versus intravenous cisplatin plus intravenous cyclophosphamide for stage III ovarian cancer. N Engl J Med. 1996 Dec 26;335(26):1950-5. doi: 10.1056/NEJM199612263352603. PMID 8960474
- [Result] Markman M, Bundy BN, Alberts DS, Fowler JM, Clark-Pearson DL, Carson LF, Wadler S, Sickel J. Phase III trial of standard-dose intravenous cisplatin plus paclitaxel versus moderately high-dose carboplatin followed by intravenous paclitaxel and intraperitoneal cisplatin in small-volume stage III ovarian carcinoma: an intergroup study of the Gynecologic Oncology Group, Southwestern Oncology Group, and Eastern Cooperative Oncology Group. J Clin Oncol. 2001 Feb 15;19(4):1001-7. doi: 10.1200/JCO.2001.19.4.1001. PMID 11181662
- [Result] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Result] Eoh KJ, Lee JY, Nam EJ, Kim S, Kim YT, Kim SW. Long-Term Survival Analysis of Intraperitoneal versus Intravenous Chemotherapy for Primary Ovarian Cancer and Comparison between Carboplatin- and Cisplatin-based Intraperitoneal Chemotherapy. J Korean Med Sci. 2017 Dec;32(12):2021-2028. doi: 10.3346/jkms.2017.32.12.2021. PMID 29115086
- [Result] Cascales-Campos P, Gil J, Feliciangeli E, Parrilla P. HIPEC in ovarian cancer: treatment of a new era or is it the end of the pipeline? Gynecol Oncol. 2015 Nov;139(2):363-8. doi: 10.1016/j.ygyno.2015.06.012. Epub 2015 Jun 16. PMID 26091936
- [Result] Trimble EL, Christian MC. Intraperitoneal chemotherapy for women with advanced epithelial ovarian carcinoma. Gynecol Oncol. 2006 Jan;100(1):3-4. doi: 10.1016/j.ygyno.2005.12.006. No abstract available. PMID 16368439
- [Result] van Driel WJ, Koole SN, Sikorska K, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AGJ, Verwaal VJ, Kieffer JM, Van de Vijver KK, van Tinteren H, Aaronson NK, Sonke GS. Hyperthermic Intraperitoneal Chemotherapy in Ovarian Cancer. N Engl J Med. 2018 Jan 18;378(3):230-240. doi: 10.1056/NEJMoa1708618. PMID 29342393
- [Result] Gouy S, Ferron G, Glehen O, Bayar A, Marchal F, Pomel C, Quenet F, Bereder JM, Le Deley MC, Morice P. Results of a multicenter phase I dose-finding trial of hyperthermic intraperitoneal cisplatin after neoadjuvant chemotherapy and complete cytoreductive surgery and followed by maintenance bevacizumab in initially unresectable ovarian cancer. Gynecol Oncol. 2016 Aug;142(2):237-42. doi: 10.1016/j.ygyno.2016.05.032. Epub 2016 Jun 2. PMID 27246305